## **Statistical Analysis**

The intention-to-treat analysis included all patients who received at least one dose of apatinib. The population assessable for treatment activity comprised all patients for whom at least one disease assessment (either clinical or radiological) was done. The primary endpoint was analysed in the intention-to-treat population. We estimated survival endpoints according to the Kaplan- Meier method, with 95% CIs. RECIST overall responses and disease control were calculated and reported with 95% CIs. We investigated the effect of P-ERK1/2 and P-RPS6 expression by comparing survival outcomes with the two-sided Mantle-Cox log-rank test, Fisher's exact test, and the Mantel-Haenszel odds ratio (OR) estimate. We compared baseline versus on-treatment PAS and BPI scores with a paired student's t test. We computed all statistics with IBM SPSS Statistics (version 20) and GraphPad Prism (version 5).